CLINICAL TRIAL: NCT05039502
Title: The Effect of Different File Systems Used in Retreatment on the Release of Inflammatory Mediators
Brief Title: Releasing of Inflammatory Mediators During Retreatment of Root Canals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sevinç Aktemur Türker, Associate Professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-27194235-01
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Response; Root Canal Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Retreatment system using in rotational motion (Experimental): Previous root canal filling materials were removed with D1-D2-D3 retreatment files with using an endodontic motor in rotational motion
  Interventions: Other: Protaper Universal Retreatment
- Retreatment system using in reciprocal motion (Experimental): Previous root canal filling materials were removed with Reciproc 25 file with using an endodontic motor in reciprocal motion
  Interventions: Other: Reciproc
- Retreatment system using in additional rotational motion (Experimental): Previous root canal filling materials were removed with XP-endo finisher r file with using an endodontic motor in rotational motion
  Interventions: Other: XP-Endo finisher R

INTERVENTIONS:
Other: Protaper Universal Retreatment — D1-D2-D3 Retreatment files were used in 500 rpm and 3 Ncm with X-Smart endomotor
  Arms: Retreatment system using in rotational motion
Other: Reciproc — R25 retratment files were used with X-Smart endomotor in reciprocal motion
  Arms: Retreatment system using in reciprocal motion
Other: XP-Endo finisher R — XP-Endo finisher r file were used in 1000 rpm 1 Ncm with X-Smart endomotor
  Arms: Retreatment system using in additional rotational motion

SUMMARY:
Nonsurgical root canal retreatment may become essential when the initial endodontic treatment fails because of the persistent intracanal or extracanal infections.The aim of this thesis study is to evaluate the effect of ProTaper Universal Retreatment (PTUR), Reciproc blue and XP-endo Finisher R file systems, which are used in the removal of root canal filling materials during retreatment with different motion kinetics on the release of Substance P, Calcitonin Gene-Related Peptide (CGRP), IL-6 and IL-10 inflammatory mediators in the periapical region

DETAILED DESCRIPTION:
Seventy-five individuals with asymptomatic and chronic apical periodontitis teeth with retreatment indication were included in the study. Individuals were randomly divided into three groups according to the file system used to remove root canal filling materials (n = 25): ProTaper Universal Retreatment, Reciproc blue and XP-endo Finisher R.After the removal of the previous root canal filling materials, reshaping and disinfection of the root canals, periapical fluid samples were taken from the root tip of the teeth in all three groups. The amount of Substance P, CGRP, IL-6 and IL-10 mediators that cause pain, swelling and flare-up in periapical fluid samples were measured by ELISA test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had single root canal treated teeth with chronic periapical lesion

Exclusion Criteria:

* Patients who are immunocompromised
* Patients under antibiotic or analgesic medication

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
change of inflammatory mediator level | 24 hours
  The samples were collected from periapical exudate at the end of the root canal retreatment procedure. The samples were analyzed with ELISA method and change of inflammatory mediator levels were evaluated in pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Sevinç Aktemur Türker, Study Director — Bulent Ecevit University
Locations (1):
- Faculty of Dentistry of Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasikci S, Turker SA, Guven B. Effect of different retreatment files using different kinematics on the release of inflammatory mediators in root canal retreatment of single-rooted teeth: a randomized clinical trial. Clin Oral Investig. 2023 Jun;27(6):3189-3196. doi: 10.1007/s00784-023-04930-6. Epub 2023 Mar 1. PMID 36856848